CLINICAL TRIAL: NCT06501365
Title: Post-Intensive Care Transitional Care, Rehabilitation, and Family-Support RCT
Brief Title: Post-Intensive Care Transitional Care, Rehabilitation, and Family-Support
Acronym: PIC-TRFS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: NOA from AHRQ never arrived, reportedly due to staffing shortages delaying grants administration. After multiple attempts to elicit a timeline from grants administration, we paused the study with hope to resume recruitment when the NOA arrives.
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Scheunemann, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY23110156; R01HS029870-01 (AHRQ)
Record Dates: First submitted 2024-07-01; First posted 2024-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care Unit Syndrome; Disabilities Multiple; Critical Illness; Caregiver Burden
Keywords: Transitional Care; Health Services; Critical Care; Post Intensive Care Unit Syndrome (PICS); Family Caregiver Support; Post Intensive Care Unit Syndrome Family (PICS - F)
MeSH Terms: conditions — Critical Illness; Caregiver Burden

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and Interventionists cannot be masked to group assignment. The Principal Investigator will remain masked. While most outcomes are patient-reported, Outcomes Assessors will be trained to remind participants not to disclose their group status during assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIC-TRFS Intervention (Experimental): Post-Intensive Care Transitions, Rehabilitation and Family Support (PIC-TRFS) is a complex dyadic intervention consisting of 4 essential elements: (1) rehabilitation; (2) health and symptom management; (3) social support; (4) healthcare coordination. It is delivered by an interventionist team. One trained interventionist leads the healthcare coordination, health and symptom management, and social support. An occupational therapist interventionist leads the rehabilitation. Following a Run-In period in the hospital, the interventionists deliver PIC-TRFS via telehealth from the time of randomization at discharge until 6 months after discharge. This Team partners with survivors, families, and the usual care team to deliver the active ingredients of PIC-TRFS.
  Interventions: Other: Post Intensive Care Transitions Rehabilitation and Family Support (PIC-TRFS)
- Enhanced Usual Care Control (Active Comparator): After receiving the Run-In and being randomized to control, this group will receive a brochure on critical illness survivorship, outcome ascertainment on the same schedule as the intervention group, and intervention for serious adverse events (e.g., suicidal ideation) identified during study conduct. This design limits exposure of the control group to the hypothesized essential elements of the PIC-TRFS intervention, while maintaining regular contact to enhance retention and outcomes ascertainment, and addressing safety concerns among participants.
  Interventions: Other: Enhanced Usual Care Control

INTERVENTIONS:
Other: Post Intensive Care Transitions Rehabilitation and Family Support (PIC-TRFS) — PIC-TRFS is a complex dyadic intervention consisting of 4 essential elements:
  1. rehabilitation;
  2. health and symptom management;
  3. social support;
  4. healthcare coordination
  It is delivered by an interventionist team via telehealth from the time of randomization at discharge until 6 months after discharge. This Team partners with survivors, families, and the usual care team to deliver the active ingredients of PIC-TRFS.
  Arms: PIC-TRFS Intervention
Other: Enhanced Usual Care Control — Dyads randomized to the Control group will receive: (1) the Run-In; (2) an informational brochure on the post-Intensive Care Syndrome; (3) ongoing assessments on the same schedule as the PIC-TRFS intervention; (4) referral for urgent emergent issues identified during the study
  Arms: Enhanced Usual Care Control

SUMMARY:
The goal of this randomized control trial is to test an intervention designed to improve patient and family outcomes after critical illness compared to usual care. The intervention, called Post-Intensive Care Transitions, Rehabilitation and Family Support (PIC-TRFS) combines four elements: (1) health management; (2) rehabilitation; (3) social support; (4) care coordination. All patients and families enrolled in this study will have spent at least 48 hours in an ICU, be at risk for long-term functional impairment, and be discharged home. Although age of the patients will be restricted to those who are at least 50 years old and caregivers must be adults over 18 and all participants must speak English, the study will enroll all sexes, genders, races, and ethnicities. The main questions the study aims to answer are:

1. Compared to usual care, does PIC-TRFS improve patient quality of life at the end of the 6-month intervention period measured via PROMIS-Preferences (PROPr) score?
2. Compared to usual care, does PIC-TRFS improve patient physical, cognitive, and psychological functioning measured via PROMIS Physical, Cognitive, and Depression Computer Adaptive Test (CAT) at 6 and 12 months after discharge? Does it increase the number of days survivors spend alive at home in the 6 and 12 months after discharge? Does it improve patient and family trauma scores and dyadic quality of life, measured via the Impact of Events Scale-Revised and dyadic PROPr score?

Participants will:

* Complete Run-In assessments of symptoms and function in the hospital;
* Be randomized to intervention or control;
* Complete assessments of their function and quality of life at 0, 3, 6 and 12 months
* Control participants will get a brochure on the Post-Intensive Care syndrome and complete the assessments on the same schedule as those receiving the intervention
* Intervention participants will complete tele-health based check-ins providing health management, social support, and care coordination; and telehealth-based rehabilitation sessions focusing on patient functioning.

DETAILED DESCRIPTION:
Each year in the United States, over 3 million people survive critical illness only to experience long-term physical, cognitive, and psychological functional impairments that contribute to ongoing health problems, high healthcare costs, and early death. Gaps in care delivery contribute to poor outcomes and preventable rehospitalizations for both patients and families. In response to these gaps, the study team used community engagement to design an intervention with 4 elements: (1) rehabilitation; (2) health and symptom management; (3) social support; (4) healthcare coordination. The result is the PIC-TRFS, which stands for Post-Intensive Care Transitional care, Rehabilitation, and Family Support (PIC-TRFS).

PIC-TRFS combines in-person and telehealth support delivered by an interdisciplinary team to nimbly address health, rehabilitation, social, and care coordination needs in collaboration with existing hospital, home health, and primary care providers. The PIC-TRFS team follows participants across transitions from hospital to home in the six months following a critical illness hospitalization. This single center randomized control trial will test whether PIC-TRFS improves outcomes compared to Enhanced Usual Care. Specifically, this research will test whether PIC-TRFS improves survivor quality of life, days alive at home, function, trauma symptoms, and family care partner quality of life. It will also test whether PIC-TRFS reduces healthcare utilization, measured as a combination of days in a healthcare facility, Emergency Department visits, and outpatient visits. At the same time, this research will assess how consistently the intervention is delivered to make sure that differences between groups really reflect the impact of the intervention. Finally, the study will explore whether the intervention may reduce health disparities between people with higher health and social needs. Successful conduct of this trial will test whether PIC-TRFS works, generate insight into how it works, and identify its impact on health equity.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet all of the following criteria:

1. All genders; Age ≥ 50
2. Admission to the hospital from home/independent living
3. Receive treatment in an ICU for ≥ 48 hours
4. At least some risk of ongoing functional impairment, measured as Activity Measures for Post-Acute Care (AMPAC) < 24, Highest Level Mobility (HLM) < 8, Intensive Care Delirium Screening Checklist (ICDSC) > 2, Significant mental health impairment (major depression, generalized anxiety, PTSD, substance use disorder)
5. Provider or e-prognosis that they are reasonably likely to be alive in 12 months (answers no to "Would you be surprised if this person were alive in 12 months?' or eprognosis risk of 1-year mortality <= 35%
6. Willingness to adhere to the PIC-TRFS regimen.
7. Provision of signed and dated informed consent form

In order to be eligible to participate in this study, a family caregiver must meet all of the following criteria:

1. All genders; Age ≥ 18 years old
2. In the survivor's social network
3. Planning to provide at least some in-home support for the survivor after discharge
4. Willingness to adhere to the PIC-TRFS regimen
5. Provision of signed and dated informed consent form

In order to be eligible for randomization, dyads must meet all of the following criteria:

1. Completion of at least the following elements of the Run-In:

   1. Patient: demographics, social needs screening tool, symptom bother scale, brief health literacy screening tool, past medical history, baseline function (Katz, Lawton, and caregiver-reported IQCODE), health priorities & goals, discharge information
   2. Caregiver: demographics, social needs screening tool, caregiver needs screening, brief health literacy screening, family caregiver training
2. Discharge to home/independent living

Exclusion criteria

Survivors will be excluded if any of the following apply:

1. They lack a family caregiver willing to participate;
2. They have a chronic condition for which they are already receiving dedicated transitional care services (e.g., post-cardiac arrest, transplant, TAVR, etc)
3. They have chronic functional dependency without potential to increase participation in meaningful activity
4. They reside outside of Pennsylvania (interventionists are only licensed to practice here)
5. They are unable to participate in English

A family caregiver who meets any of the following criteria will be excluded from participation in this study:

1. They are unable to participate in English

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in mean patient PROMIS-Preferences at the end of the intervention period | 6 months
  Patients will report health-related quality of life using Patient Reported Outcomes Measurement Information System (PROMIS) surveys in 7 domains: physical, cognitive, mental health, social role satisfaction, pain, fatigue, and sleep. The statistician will use the surveys to calculate a PROMIS-Preferences (PROPr) score using the code available here https://www.proprscore.com/code-and-data/ . This yields a T-score with a minimum of -0.022 (worse than dead) and a maximum score of 1 (maximum quality of life). These scores will be aggregated by calculating the mean for each study group.

SECONDARY OUTCOMES:
Between-group difference in patient PROMIS-Preferences scores at the end of the study period | 12 months
  Patients will report health-related quality of life using PROMIS surveys in 7 domains: physical, cognitive, mental health, social role satisfaction, pain, fatigue, and sleep. The statistician will use the surveys to calculate a PROPr score using the code available here https://www.proprscore.com/code-and-data/ . This yields a T-score with a minimum of -0.022 (worse than dead) and a maximum score of 1 (maximum quality of life). These scores will be aggregated by calculating the mean for each study group.
Between group differences in survivor physical function | 6 and 12 months
  Patients will complete the PROMIS Physical Function Computer Adaptive Test (CAT) survey. This yields a T-score with a mean score of 50 and SD of 10, with scores of 0 representing the worst possible physical function and scores of 100 the best possible physical function. Means for each study group will be compared.
Between group differences in survivor cognitive function | 6 and 12 months
  Patients will complete the PROMIS Cognitive Function Computer Adaptive Test (CAT) survey. This yields a T-score with a mean score of 50 and SD of 10, with scores of 0 representing the worst possible cognitive function and scores of 100 the best possible cognitive function. Means for each study group will be compared.
Between group differences in survivor mood | 6 and 12 months
  Patients will complete the PROMIS Mood (Depression) CAT survey. This yields a T-score with a mean score of 50 and SD of 10, with scores of 0 representing the worst possible mood function and scores of 100 the best possible mood. Means for each study group will be compared.
Between-group differences in mean dyadic PROMIS-Preferences (PROPr) Scores | 6 and 12 months
  Patients and families will report health-related quality of life using PROMIS surveys in 7 domains: physical, cognitive, mental health, social role satisfaction, pain, fatigue, and sleep. The statistician will use the surveys to calculate a PROPr score using the code available here https://www.proprscore.com/code-and-data/ . This yields a T-score with a minimum of -0.022 (worse than dead) and a maximum score of 1 (maximum quality of life). These scores will be aggregated by adding the values of each patient-family dyad and then calculating the mean for each study group.
Between group differences in dyadic trauma symptoms | 6 and 12 months
  Patients and families will complete the Impact of Events Scale-Revised. Individual scores range from 0-88, with scores >=24 indicating clinical concern for Post Traumatic Stress Disorder (PTSD), scores >=33 indicating probably PTSD, and scores >=37 indicating severe PTSD. The statistician will sum the scores of the patient-family dyad. Assuming a normal distribution, they will compare means for each study group.
Between group differences in survivor days alive at home. | 6 and 12 months
  Survivor days alive at home at home will be measured from the time of discharge to the specified time point (6 and 12 months) post discharge. Family, primary care provider, or death certificate will confirm date of death. Days in a healthcare facility (Emergency Department, hospital or skilled nursing facility) will be self-reported via an Event Calendar. Days alive at home will be calculated by subtracting the sum of days in a healthcare facility and days dead over 6 and 12 months after discharge, respectively. Medians for each study group will be compared. Minimum value is 0 (readmitted or died on the day of discharge) and maximum is 365 (survived the year without readmission).
Between group differences in survivor Healthcare Utilization | 6 and 12 months
  Healthcare facility days and Emergency Department visits, both individually and collectively, will be extracted from: (a) patient and family report via event calendar; (b) medical record review. The statistician will sum the number of healthcare facility days and Emergency Department visits. Medians for each study group will be compared. Minimum value is 0 (no healthcare utilization, probably an indicator of extremely poor health or lack of access); a low number utilized is consistent with stable health with access (~1-12); while high utilization (>12) likely indicates unstable health with consequently high needs

CONTACTS AND LOCATIONS:
Overall Officials: Leslie P Scheunemann, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC/University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Scientific data that will be preserved and shared are demographical data and medical history. In addition, we will preserve and share self-report data obtained from critical illness survivors and caregivers, and those related to intervention delivery, receipt and enactment. Case report forms used to collect construct the EDC will be preserved and shared. Some data will be extracted from participants' electronic health records. We will also share the data dictionary and codebook.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be retained for at least 7 years after publication of the results, per institutional policy. The data will be available for sharing during this period.
Access Criteria: Those willing to access the data should initiate request to the Principal Investigator (PI) Dr. Leslie Scheunemann via email. The PI will discuss the request, purpose and merits with the team of co-investigators, collaborators and consultants. Only de-identified data will be shared. The data will be shared only after an appropriate data use agreement. Once approved, data will be transferred via email or a cloud storage platform such as OneDrive.

REFERENCES:
- [Background] Scheunemann LP, Motter EM, Kim SP, Eisenhauer P, Gandhi N, Eaton TL, Girard TD, Reynolds CF, Leland NE. Re-engineering Transitional Care After Critical Illness: A Qualitative Integration of Multiple Perspectives. Under review, 2024.
- [Background] Moale AC, Motter EM, Eisenhauer P, Gandhi N, Kim SP, Girard TD, Reynolds CF 3rd, Leland NE, Chang JC, Scheunemann LP. Integrating Perspectives on Family Caregiving After Critical Illness: A Qualitative Content Analysis. Am J Crit Care. 2024 May 1;33(3):180-189. doi: 10.4037/ajcc2024309. PMID 38688852
- [Background] Scheunemann LP, White JS, Prinjha S, Hamm ME, Girard TD, Skidmore ER, Reynolds CF 3rd, Leland NE. Post-Intensive Care Unit Care. A Qualitative Analysis of Patient Priorities and Implications for Redesign. Ann Am Thorac Soc. 2020 Feb;17(2):221-228. doi: 10.1513/AnnalsATS.201904-332OC. PMID 31726016
- [Background] Naylor MD, Hirschman KB, Toles MP, Jarrin OF, Shaid E, Pauly MV. Adaptations of the evidence-based Transitional Care Model in the U.S. Soc Sci Med. 2018 Sep;213:28-36. doi: 10.1016/j.socscimed.2018.07.023. Epub 2018 Jul 17. PMID 30055423
- [Background] Scheunemann L, White JS, Prinjha S, Eaton TL, Hamm M, Girard TD, Reynolds C, Leland N, Skidmore ER. Barriers and facilitators to resuming meaningful daily activities among critical illness survivors in the UK: a qualitative content analysis. BMJ Open. 2022 Apr 26;12(4):e050592. doi: 10.1136/bmjopen-2021-050592. PMID 35473739
- [Background] Skidmore ER, Butters M, Whyte E, Grattan E, Shen J, Terhorst L. Guided Training Relative to Direct Skill Training for Individuals With Cognitive Impairments After Stroke: A Pilot Randomized Trial. Arch Phys Med Rehabil. 2017 Apr;98(4):673-680. doi: 10.1016/j.apmr.2016.10.004. Epub 2016 Oct 26. PMID 27794487
- [Background] Skidmore ER, Swafford M, Juengst SB, Terhorst L. Self-Awareness and Recovery of Independence With Strategy Training. Am J Occup Ther. 2018 Jan/Feb;72(1):7201345010p1-7201345010p5. doi: 10.5014/ajot.2018.023556. PMID 29280726
- [Background] Rouch S, Skidmore ER. Examining Guided and Directed Cues in Strategy Training and Usual Rehabilitation. OTJR (Thorofare N J). 2018 Jul;38(3):151-156. doi: 10.1177/1539449218758618. Epub 2018 Feb 15. PMID 29444624
- [Background] Campbell GB, Boisen MM, Hand LC, Lee YJ, Lersch N, Roberge MC, Suchonic B, Thomas TH, Donovan HS. Integrating Family Caregiver Support Into a Gynecologic Oncology Practice: An ASCO Quality Training Program Project. JCO Oncol Pract. 2020 Mar;16(3):e264-e270. doi: 10.1200/JOP.19.00409. Epub 2019 Sep 7. PMID 31496394
- [Background] Hand LC, Thomas TH, Belcher S, Campbell G, Lee YJ, Roberge M, Donovan HS. Defining Essential Elements of Caregiver Support in Gynecologic Cancers Using the Modified Delphi Method. J Oncol Pract. 2019 Apr;15(4):e369-e381. doi: 10.1200/JOP.18.00420. Epub 2019 Mar 8. PMID 30849004
- [Background] Chi Y, Thaker K, He D, Hui V, Donovan H, Brusilovsky P, Lee YJ. Knowledge Acquisition and Social Support in Online Health Communities: Analysis of an Online Ovarian Cancer Community. JMIR Cancer. 2022 Sep 13;8(3):e39643. doi: 10.2196/39643. PMID 36099015
- See also: Website intended to highlight research and provide a "living toolkit" to survivors and families. — https://picturethis.pitt.edu/

DOCUMENTS (1):
  • Informed Consent Form (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT06501365/ICF_002.pdf